CLINICAL TRIAL: NCT06270498
Title: Effect of Oral sucRosomIal Iron on exerciSE Capacity and Quality of Life in Patients With Heart Failure: a Randomized, Placebo-controlled Trial (RISE-HF)
Brief Title: Effect of Oral sucRosomIal Iron on exerciSE Capacity and Quality of Life in Patients With Heart Failure
Acronym: RISE-HF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Raffaele De Caterina (Other)
Collaborators: University of Pisa (Other)
Responsible Party: Sponsor-Investigator, Raffaele De Caterina, Chair of Cardiology Division, Azienda Ospedaliero, Universitaria Pisana
Organization: Azienda Ospedaliero, Universitaria Pisana (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24811
Record Dates: First submitted 2024-02-10; First posted 2024-02-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Heart Failure; Iron-deficiency; Left Ventricular Systolic Dysfunction
Keywords: heart failure; iron deficiency; sucrosomial iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Ventricular Dysfunction, Left; Heart Failure; Iron Deficiencies | interventions — sucrosomial iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sucrosomial iron (Active Comparator)
  Interventions: Dietary Supplement: Sucrosomial iron
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sucrosomial iron — Sucrosomial iron with the addition at a fixed dose of vitamin C to promote iron absorption (SiderAL® Forte) will be administered orally once a day for 24 weeks.
  The dose regimen for all participants will be calculated according to the haemoglobin (Hb) levels at baseline evaluation and to patient's body weight as follows:
  Hb 14-16 g/dL: 1 tablet once a day, corresponding to 30 mg/daily, for 24 weeks; Hb 10-13.9 g/dL: 2 tablets once a day, corresponding to 60 mg/daily, for 24 weeks
  Other Names: SiderAL Forte
  Arms: Sucrosomial iron
Other: Placebo — Placebo pills will be identical in shape, form and color of SI tablets; they will contain the same components of SiderAL Forte® except for sucrosomial iron and vitamin C.
  Placebo will be administered orally once a day for 3 months according to the same dose scheme in the intervention arm.
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate the effect of oral sucrosomial iron on exercise capacity and quality of life in patients with heart failure (HF) and iron deficiency (ID).

The main question the study aims to answer is whether oral sucrosomial iron improved exercise capacity, assessed by six-minute walk test, and quality of life, assessed by Kansas City Cardiomyopathy Questionnaire, compared with placebo.

One group of participants will receive treatment with oral sucrosomial iron and the other group will receive treatment with placebo.

DETAILED DESCRIPTION:
Based on clinical trials, treatment with intravenous iron improves symptoms, exercise capacity, and may reduce HF hospitalizations in patients with HF and ID. On the contrary, treatment of ID with oral iron has no effect on exercise capacity. High hepcidin levels prevent oral intestinal absorption and blunt the response to oral iron administration. Sucrosomial iron (SI) consists of a nucleus of ferric pyrophosphate with an envelope of sucrose ester of fatty acids, which promotes intestinal absorption through paracellular and lymphatic routes, independent of hepcidin. In contrast with intravenous iron infusion, administration of oral iron may not promote oxidative stress, since the intestinal iron absorption prevent the formation of labile, non-transferrin bound, plasma iron.

The study will investigate the effect of oral SI supplementation on exercise capacity, assessed by six-minute walk test, and quality of life, assessed by Kansas City Cardiomyopathy Questionnaire, compared with placebo in patients with HF, a left ventricular ejection fraction (LVEF) <50%. Iron deficiency was defined as transferrin saturation (TSAT) <20%.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HF (New York Heart Association [NYHA] functional class II-IV) patients, on optimal therapy, and clinically stable for at least 4 weeks with no dose changes of HF drugs
2. LVEF<50% at screening visit (historical value can be used if performed within 6 months of screening visit)
3. Either a documented hospitalization for HF in the previous 12 months of enrolment or an elevated NT-proBNP: ≥250 pg/mL (or BNP ≥75 pg/mL) for patients in normal sinus rhythm; ≥1,000 pg/mL (or BNP ≥400 pg/mL) for patients in atrial fibrillation
4. TSAT <20%
5. Hemoglobin 10.0-16.0 g/dL
6. Rapid iron repletion with intravenous iron is not considered a clinical necessity by physicians after reviewing patient medical record (if anaemia is present, its grade is no more than mild)
7. Age ≥18 years, male and female
8. Willingness to provide informed consent
9. Subjects who decide to use single or dual contraceptive methods to avoid conceiving during the study period

Exclusion Criteria:

1. Neuromuscular, orthopedic or other non-cardiac condition that prevents the patient from exercise testing
2. Exercise training program in the previous 3 months, or planned in the next 3 months
3. Recent (<3 month) acute coronary syndrome, coronary artery bypass surgery, percutaneous coronary interventions, transient ischemic attack, or stroke
4. Severe valvular disease, hypertrophic obstructive cardiomyopathy, restrictive or constrictive cardiomyopathy, acute myocarditis
5. Atrial fibrillation or flutter with a ventricular response rate of >100 beats per minute at rest
6. Temperature ≤38 °C (oral or equivalent) or active infection as defined by current use of oral or intravenous antimicrobial agents
7. Need for blood transfusion within the last month
8. Hb<10 g/dL or Hb>16 g/dL
9. Rapid iron repletion with intravenous iron is considered a clinical necessity by physicians after reviewing patient medical record
10. Documented active gastrointestinal bleeding
11. Oral iron, i.v. iron or erythropoietin stimulating agent within the last 3 months
12. eGFR ≤15 mL/min or on hemodialysis
13. Chronic liver disease and/or alanine transaminase or aspartate transaminase above 3 times the upper limit of the normal range
14. Active cancer
15. Evidence of iron overload (ferritin >400 ng/mL)
16. Hypersensitivity to any of the study products or known severe allergies
17. Participation in another study
18. Low body weight (≤35 kg)
19. Known or anticipated pregnancy in the next 4 months
20. Need for forbidden medications
21. Breastfeeding
22. Consumption of iron-rich foods or any food that alter iron absorption (i.e. food rich in vitamin C) due to dietary requirements
23. Any pathological condition or disease associated with a reduction or an impairment of intestinal iron absorption (i.e., prior gastrectomy, atrophic gastritis, bariatric surgery, coeliac disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Difference in six-minute walk test (6MWT) distance, expressed as meters | 12 weeks
Difference in Kansan City Cardiomyopathy Questionnaire (KCCQ)-12 overall score | 12 weeks

SECONDARY OUTCOMES:
Proportion of patients with 15 meters improvement in 6MWT distance (responders) | 12 weeks
Proportion of patients with 5-point improvement in KCCQ-12 score (responders) | 12 weeks
Difference in six-minute walk test (6MWT) distance, expressed as meters | 24 weeks
Difference in Kansan City Cardiomyopathy Questionnaire (KCCQ)-12 overall score | 24 weeks
Proportion of patients with 15 meters improvement in 6MWT distance (responders) | 24 weeks
Proportion of patients with 5-point improvement in KCCQ-12 score (responders) | 24 weeks
Bone metabolism indices | 12 weeks
  Change in phosphate and FGF-23
Bone metabolism indices | 24 weeks
  Change in phosphate and FGF-23
Iron indices | 12 weeks
  Change in TSAT, ferritin and serum iron
Iron indices | 24 weeks
  Change in TSAT, ferritin and serum iron
Oxidative stress | 12 weeks
  Change in F2-isoprostanes, Soluble NOX2-derived peptide and H2O2
Oxidative stress | 24 weeks
  Change in F2-isoprostanes, Soluble NOX2-derived peptide and H2O2
Iron indices 2 | 12 weeks
  change in soluble receptor of transferrin and hepcidin
Iron indices 2 | 24 weeks
  change in soluble receptor of transferrin and hepcidin
Systolic cardiac function | 12 weeks
  Change in Left ventricular ejection fraction, %
Systolic cardiac function | 24 weeks
  Change in left ventricular ejection fraction, %
NTproBNP | 12 weeks
  Change in NT-proBNP
NTproBNP | 24 weeks
  Change in NT-proBNP
Clinical events | 12 weeks
  Time to death or to first HF hospitalization
Clinical events | 24 weeks
  Time to death or to first HF hospitalization
Left atrial volume | 12 weeks
  Change in left atrial volume
Left ventricular volume | 12 weeks
  Change in left ventricular end-diastolic volume
Left ventricular diastolic function | 12 weeks
  change in E/e' ratio
Echocardiographic estimation of pulmonary pressure | 12 weeks
  change in systolic pulmonary artery pressure
Left atrial volume | 24 weeks
  Change in left atrial volume
Left ventricular diastolic function | 24 weeks
  change in E/e' ratio
Echocardiographic estimation of pulmonary pressure | 24 weeks
  change in systolic pulmonary artery pressure
Left ventricular volume | 24 weeks
  Change in left ventricular end-diastolic volume

OTHER OUTCOMES:
Adverse events and allergic reactions | 12 weeks
  Number of any adverse events and number of allergic reactions
Adverse events and allergic reactions | 24 weeks
  Number of any adverse events and number of allergic reactions

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Masini, MD PhD, Principal Investigator — University of Pisa; Raffaele De Caterina, MD PhD, Study Director — University of Pisa
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: Undecided